CLINICAL TRIAL: NCT03535259
Title: Phase II Study of Concurrent Sorafenib and Intensity-modulated Radiotherapy (IMRT) for Advanced Hepatocellular Carcinoma
Acronym: SIRAHCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, BO CHEN, Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC201803020
Record Dates: First submitted 2018-05-12; First posted 2018-05-24 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma, Radiotherapy, Sorafenib
Keywords: hepatocellular carcinoma; intensity-modulated radiotherapy; sorafenib; portal vein thrombosis; lymph node metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Lymphatic Metastasis | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sorafenib and IMRT (Experimental): Concurrent sorafenib and IMRT, followed sorafenib maintenance for advanced hepatocellular carcinoma with portal vein or hepatic vein tumor thrombosis or lymph node involved
  Interventions: Radiation: concurrent sorafenib and IMRT, followed sorafenib maintenance

INTERVENTIONS:
Radiation: concurrent sorafenib and IMRT, followed sorafenib maintenance — IMRT 40-60Gy/20-30f; concurrent sorafenib 400mg bid po (it can be given to patients in four weeks before IMRT is applied, so that it can control disease during waiting for IMRT); maintenance sorafenib 400mg bid po until disease progress or unacceptable adverse events; six months is recommended but not mandatory.

SUMMARY:
This is a single-arm phase II clinical trial to investigate the efficacy and toxicity of concurrent sorafenib and intensity-modulated radiotherapy (IMRT) for advanced hepatocellular carcinoma with portal vein or hepatic vein tumor thrombosis or lymph node involved. Eligibility patients will receive IMRT to hepatic primary tumor, vein tumor thrombosis, and metastasis lymph node with concurrently sorafenib with a dose of 400mg twice daily. Prescription of IMRT will be a conventional fraction dose of 2Gy to a total dose of 40 to 60Gy. Sorafenib will be maintained with a dose of 400mg twice daily after IMRT until disease progression, or unacceptable adverse events. Six months of sorafenib maintenance is recommended.

DETAILED DESCRIPTION:
With the clinical application of three-dimensional conformal radiotherapy (3DCRT) and intensity modulated radiotherapy (IMRT), radiotherapy (RT) has shown important role in the treatment of hepatocellular carcinoma (HCC). Meta-analysis has demonstrated that transcatheter arterial chemoembolization (TACE) combined RT was more therapeutically beneficial than TACE alone. Especially for advanced disease with portal vein tumor thrombosis (PVTT), or hepatic vein tumor thrombosis, or lymph node involved, RT was more effective than other treatment methods. Previous studies had showed that RT could receive response rate of 50% to 60% for HCC with PVTT. But for those patients, high accidence of out RT field failure of liver and distance metastasis was found. Effective systemic therapy was necessary to advanced HCC. Based on two phase III trials, sorafenib was recommended as systemic therapy to advanced HCC. But tumor response rate of sorafenib alone was only 2.3-3% by RICIST criteria. More than half of patients was received survival benefit by maintaining in stable disease. It is feasible to improve survival by combining IMRT and sorafenib for advanced HCC with portal vein tumor thrombosis (PVTT), or hepatic vein tumor thrombosis, or lymph node involved. In addition, it was demonstrated that sorafenib could potentiate irradiation in HCC cell lines through inhibiting radiation-induced proliferation and DNA repair and promoting radiation-induced apoptosis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical or histologic diagnosis of Hepatocellular carcinoma (HCC)
2. Aged between 18 and 80 years
3. ECOG 0-1
4. Liver-GTV>700ml
5. BCLC stage C, HCC with portal vein or hepatic vein tumor thrombosis or lymph node involved (LN involved can be included one treatment planning)
6. Estimated life expectancy > 3 months
7. Child-Pugh Score: A5-B8
8. Hepatic function: alanine transaminase (ALT) and aspartate transaminase (AST)≤ 1.5 times ULN; or ALT ≤ ULN and AST≤ 6 times ULN exclude possibility of heart disease
9. Renal function: creatinine (CRE) and blood urea nitrogen (BUN)≤ 1.5 times ULN
10. Blood routine examination: Hb≥80g/L, ANC≥1.0×109 /L, PLT≥40×109 /L
11. Voluntary to participate and sign informed consent

Exclusion Criteria:

1. Had prior abdominal irradiation
2. Had prior liver transplantation
3. Had serious myocardial disease or renal failure
4. Pregnant, breast feeding, or unwilling to use adequate contraception
5. Known hypersensitivity to sorafenib

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
MST | 24 months
  Median Survival Time (MST) was defined as the duration from the date of patient recruited to the date of death from any cause

SECONDARY OUTCOMES:
ORR | Assessment in 1 to 3 months after IMRT
  Overall Response Rate (ORR) was defined as the total of CR (Complete Response) and PR (Partial Response). CR and PR were assessed by independent reviewers according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. ORR evaluated in 1 to 3 months after the completion of IMRT.
TTP | 24 months
  Time to Progression (TTP) was defined as the duration from the date of patient recruited to the first progress at any site or the date of death
Rate of III-IV grade adverse events | up to 24 months
  Adverse events was evaluated during received protocol therapy according to CTCAE 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Bo Chen, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhai Y, Wang L, Zhao H, Wu F, Xin L, Ye F, Sun W, Song Y, Niu L, Zeng H, Wang J, Tang Y, Song Y, Liu Y, Fang H, Lu N, Jing H, Qi S, Zhang W, Wang S, Li YX, Wu J, Chen B. Phase II study with sorafenib plus radiotherapy for advanced HCC with portal and/or hepatic vein tumor thrombosis. JHEP Rep. 2024 Nov 28;7(3):101287. doi: 10.1016/j.jhepr.2024.101287. eCollection 2025 Mar. PMID 39980754